CLINICAL TRIAL: NCT06693700
Title: Freedom to Breathe: Pilot Study Towards Achieving Environmental Justice for Cancer Patients and Their Families
Brief Title: A Study Evaluating the Use of an Indoor Air Quality Monitor to Promote a Smoke-free Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-260
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Smoking; Smoking Cessation; Smoking Reduction; Smoking Habit; Smoking Behaviors; Smoking, Tobacco; Smoking, Cigarette; Smoking (Tobacco) Addiction; Tobacco Use; Tobacco Smoking
Keywords: smoking; smoking cessation; smoking reduction; smoking habit; smoking behaviors; smoking, tobacco; smoking, cigarette; smoking (tobacco) addiction; tobacco use; tobacco smoking; air quality; indoor air quality monitoring devices; 24-260; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Smoking; Smoking Cessation; Smoking Reduction; Tobacco Smoking; Cigarette Smoking; Behavior, Addictive; Tobacco Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSK Participants who are current smokers (Experimental): 10 MSK participants who are current smokers and receiving tobacco treatment will be enrolled.
  Interventions: Other: Indoor Air Quality Monitor AirGradient ONE

INTERVENTIONS:
Other: Indoor Air Quality Monitor AirGradient ONE — Participants will be asked to set up an Indoor Air Quality Monitor AirGradient ONE (Model: I-9PSL) which is an award winning commercially available indoor air quality monitor designed to enable anyone to monitor their air quality in their home for about 60 days (8 weeks). Indoor air pollution levels within participating households will be measured using these AQMs.

SUMMARY:
The purpose of this study is to evaluate how using an indoor air quality monitor can promote a smoke-free home for cancer patients who are enrolled in MSK's Tobacco Treatment Program.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged >18 years) MSK patients as per the EHR
* Has been referred and enrolled in the MSK TTP and completed the initial counseling session as per the TTP clinical database
* Reports current (within the past 30 days) tobacco use (i.e., cigarettes and/or any other tobacco products) as per the TTP Intake form
* Must be English-speaking in the EHR
* Must be reachable by phone as per self-report
* Must have Wi-Fi available at home as per self-report

Exclusion Criteria:

* Patient reports that no smoking is allowed, by them or anyone else, in the home as per the TTP intake form and/or per self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-11-14 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants using the air quality monitoring device for 14 consecutive days | up to 8 weeks
  Assess the feasibility and acceptability of collecting environmental data on biomarkers of household air quality (AQ) and smoke exposure using low-cost, AQMs as an intermediate endpoint of a smoke-free-home.
Percentage of participants who attend the study-specific smoke-free workshop sessions | Up to 8 weeks
  Assess the feasibility and acceptability of tobacco treatment adherence among individuals diagnosed with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Gleneara Bates-Pappas, PhD, LMSW, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - City College of New York (Data Collection AND Data Analysis), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org